CLINICAL TRIAL: NCT05085795
Title: Impulse Oscillometry and the Bronchoprotective Effects of Deep Inspiration
Brief Title: Evaluating Deep Breathing in Health Participants Using a Device Called Impulse Oscillometry
Status: Completed | Type: Observational
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Steve Nicholas Georas, Professor, University of Rochester
Other Study IDs: STUDY00006488
Record Dates: First submitted 2021-10-07; First posted 2021-10-20 (Actual); Last update posted 2023-08-15 (Actual); Status verified 2023-08

CONDITIONS: Breathing, Mouth; Lung Function Decreased
MeSH Terms: conditions — Mouth Breathing; Respiratory Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- All participants
  Interventions: Device: Impulse Oscillometer

INTERVENTIONS:
Device: Impulse Oscillometer — The tremoFlo C-100 Airwave Oscillometry System is intended to measure respiratory system impedance using the Forced Oscillation Technique (FOT).
  Other Names: THORASYS tremoFlo C-100 Airwave Oscillometry System

SUMMARY:
This study will determine if resistance of the airway to airflow and pressure, measured by Impulse Oscillometry, is impacted by a deep breathe maneuver in a small cohort of healthy human subjects.

ELIGIBILITY:
Inclusion Criteria:

* Vaccinated against COVID-19
* Ability to provide informed consent
* Willingness to perform breathing test
* Willingness to provide basic demographic data
* Must be able to speak and understand English

Exclusion Criteria:

* Unable to or unwilling to provide consent, perform test, or provide basic demographic data

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Up to fifty (50) healthy subjects will be recruited from Mary Parkes Asthma and Allergy Center and the outpatient pulmonary clinics at the University of Rochester Medical Center, and from the Pulmonary and Critical Care Division at the University of Rochester
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2021-10-04 (Actual); Primary Completion 2022-05-27 (Actual); Study Completion 2023-08-08 (Actual)

PRIMARY OUTCOMES:
Mean respiratory system impedance | pre deep inspiration, approximately day 1
  The oscillometer will collect an airway impedance measurement which is made up of multiple variables.
Mean respiratory system resistance | post deep inspiration, approximately day 1
  The oscillometer will collect an airway impedance measurement which is made up of multiple variables.
Mean change in respiratory system resistance | post and pre deep inspiration, approximately day 1
  The oscillometer will collect an airway impedance measurement which is made up of multiple variables.

CONTACTS AND LOCATIONS:
Locations (1):
- Mary Parkes Asthma and Allergy Center, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (2):
  • Study Protocol (2022-02-14): https://cdn.clinicaltrials.gov/large-docs/95/NCT05085795/Prot_000.pdf
  • Informed Consent Form (2022-02-15): https://cdn.clinicaltrials.gov/large-docs/95/NCT05085795/ICF_001.pdf